CLINICAL TRIAL: NCT07147894
Title: Understanding Mediating and Moderating Factors That Determine Transfer of Working Memory Training in Adolescents
Brief Title: Executive Function Training for Children and Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NU-23-05-12
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Cognitive Change
Keywords: ADHD; Executive Function Training; Motivational coaching; Cognitive Training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one out of six training conditions. The training conditions are as follows: (1) Nongamified n-Back; (2) Gamified n-Back; (3) Multiple Domain Training; (4) Nongamified n-Back + Motivational Coaching; (5) Gamified n-Back + Motivational Coaching; (6) Multiple Domain Training + Motivational Coaching
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Non Gamified N-back Training (Experimental): Participants train on a non gamified version of the N-back task.
  Interventions: Behavioral: Nongamified N-back training
- Gamified N-back Training (Experimental): Participants train on a gamified version of the N-back task.
  Interventions: Behavioral: Gamified N-back training
- Multiple Domain Training (Experimental): Participants train on N-Back, Complex Span, Set Shifting (Polyrules), and Inhibitory Control.
  Interventions: Behavioral: Multiple Domain Training
- Non Gamified N-back Training with Coaching (Experimental): Participants train on a non gamified version of the N-Back task and will receive weekly, motivational coaching sessions via videoconference.
  Interventions: Behavioral: Nongamified N-back training; Behavioral: Coaching Session
- Gamified N-back Training with Coaching (Experimental): Participants train on a gamified version of the N-back task and will receive weekly, motivational coaching sessions via videoconference.
  Interventions: Behavioral: Gamified N-back training; Behavioral: Coaching Session
- Multiple Domain Training with Coaching (Experimental): Participants train on gamified N-back training, Complex Span, Set Shifting, and Inhibitory Control and also receive weekly, motivational coaching sessions via videoconference.
  Interventions: Behavioral: Multiple Domain Training; Behavioral: Coaching Session

INTERVENTIONS:
Behavioral: Nongamified N-back training — This Single Task Training is an adaptive N-back task in which participants respond to colors and/or shapes.
  Arms: Non Gamified N-back Training
Behavioral: Gamified N-back training — Participants train on a gamified version of the N-back task, specifically, players control an astronaut that collects resources (target stimuli) needed to feed a colony and keep the technology working, while avoiding non-targets and other obstacles.
  Arms: Gamified N-back Training; Gamified N-back Training with Coaching
Behavioral: Multiple Domain Training — Participants train on a gamified versions of the N-back task, Complex span, Set-shifting and Inhibitory control task.
  Arms: Multiple Domain Training; Multiple Domain Training with Coaching
Behavioral: Nongamified N-back training — This Single Task Training trains a visual, adaptive N-back task in which participants respond to colors and/or shapes.
  Arms: Non Gamified N-back Training with Coaching
Behavioral: Coaching Session — Participants in coaching conditions receive weekly, motivational coaching sessions via videoconference to (i) provide encouragement taking into account individual training performance and self-reported engagement (strength-based feedback), (ii) set realistic goals for training (time management, scheduling, and session completion plan, performance goals) while emphasizing autonomy and choice, and (iii) re-explain task and provide corrective feedback as needed.
  Arms: Gamified N-back Training with Coaching; Multiple Domain Training with Coaching; Non Gamified N-back Training with Coaching

SUMMARY:
The goal of this clinical trial is to evaluate how different approaches to executive function (like adding game-like features, varying the number of tasks, and providing coaching) can enhance executive function outcomes in adolescents with and without ADHD. The main questions it aims to answer are:

* What components of executive function training contribute most to improving outcomes?
* How do training components vary in their impacts on adolescents diagnosed with ADHD compared to those without a diagnosis?
* What individual characteristics influence the effectiveness of executive function training?

Researchers will test six different training setups to examine which setups are the most effective for different people. They will evaluate both how well participants follow the training schedule and whether there are changes in psychological and cognitive outcomes after training.

Participants will complete:

* 40 training sessions over 4 weeks
* A set of tests and surveys before and after the training
* Follow-up assessments and surveys 6 months after finishing the training

ELIGIBILITY:
Inclusion Criteria:

* 12-17 years old.
* Child must have a caregiver (parent/guardian) who is available to participate as a training aide.
* Child and parent/caregiver are able to understand/speak adequate English or Spanish to follow and participate in study procedures
* Both child and parent/guardian are willing to give informed consent/assent, be randomized to either intervention condition, and be willing to follow the assigned study protocol.
* ~50% of the participants: Meet criteria for ADHD DSM-5 diagnosis.

Exclusion Criteria:

* Child is taking ADHD medication/stimulants.
* Child has been formally identified as intellectually disabled.
* Abnormal visual acuity or hearing challenges that are prohibitive to participating in the intervention/assessment.
* History of organic mental disorders (conditions or disturbances that may be caused by injuries and/or neurodegenerative diseases affecting brain tissues), psychosis, history of autism spectrum disorders, intellectual disability, or active substance use or suicidal ideation (such individuals will be referred to psychiatric services).
* Major sensory or motor impairment that would preclude valid cognitive testing.
* Participants with color blindness, if they are unable to discriminate the task relevant stimuli.
* Populations considered vulnerable such as wards and those with neurological or other health conditions that may prevent the ability to give informed consent.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 780 (Estimated)
Dates: Start 2025-12-14 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Adherence Composite | 40 training sessions (weeks 2-5)
  An Adherence Composite will be an aggregate score between (1) Participant compliance assessed by the number of completed training sessions completed within guidelines. For each completed training session that complies with the schedule, participants will receive one point, for a total of 40 possible points; (2) Self-reported engagement: After each training session, children are asked to rate their level of engagement using a Likert scale. The dependent variable will be the average engagement rating across all completed sessions; and (3) Effort, which is assessed by fitting a curve to daily training performance with 1 point given for each session where performance is at or above 0.5 SD of the daily estimate for a total of 40 possible points. Furthermore, after each training session, children are asked to rate their level of effort put into the training using a visualized Likert scale. All adherence measures will be combined across all the measures to compute a composite score.
Working Memory Composite | pre-test (week 1), post-test (week 6), and 1 follow-up session at least 6 months after post-test (week 30).
  A composite score across 3 working memory measures will be computed. (1) Spatial working memory span is a game-like version of the Corsi-blocks task to assess visuospatial working memory; dependent variable: maximum span length. (2) Complex working memory span is similar to Spatial working memory span but also includes a sorting task in-between encoding trials; dependent variable: maximum span length. In (3) Letter-Number Sequencing, participants are presented with a series of intermixed stimuli (e.g., letters and numbers) and recall each stimulus category separately in numerical/alphabetical order; dependent variable: maximum span length.
Inhibition/Flexibility Composite | pre-test (week 1), post-test (week 6), and 1 follow-up session at least 6 months after post-test (week 30).
  A composite score across inhibitory control/set-shifting measures will be computed. (1) Continuous performance task, modeled after standard measures; dependent variable: hits minus false alarms. (2) Flanker task: classic flanker task; dependent variable: a score based upon speed and accuracy. (3) Rule Switch task a standard switching task; dependent variable: is a score based upon speed and accuracy.

SECONDARY OUTCOMES:
Complex Cognition Composite | pre-test (week 1), post-test (week 6), and 1 follow-up session at least 6 months after post-test (week 30).
  A composite across the following measures will be computed. (1) Fluid Intelligence will be measured with the UCMRT matrix reasoning task; dependent variable: number of correct responses. (2) Quantitative Skills will be assessed through a basic arithmetic task where participants quickly answer addition, subtraction multiplication, and division questions; dependent variable: number of correct responses. Finally, we test (3) Reading Speed will be assessed through a basic where short stories are read, and participants answer comprehension at the end of each passage; dependent variable: composite score of time to complete the task and number of correct responses.
Well-Being Composite | pre-test (week 1), post-test (week 6), and 1 follow-up session at least 6 months after post-test (week 30).
  A composite score across standardized surveys to assess self-perceived stress and quality of life will be used.
Mental Health Composite | pre-test (week 1), post-test (week 6), and 1 follow-up session at least 6 months after post-test (week 30).
  A composite across standardized surveys that capture ADHD symptoms will be used across the full sample; in addition, we will assess functional outcomes in the ADHD sample.

OTHER OUTCOMES:
Control Measures | pre-test (week 1), post-test (week 6), and 1 follow-up session at least 6 months after post-test (week 30).
  We will also examine measures that we do not expect to change. Vocabulary and General Knowledge will be assessed using standardized tests that require participants to select the appropriate response among several alternatives. Dependent variable: number of correct responses.
Near Transfer | pre-test (week 1), post-test (week 6), and 1 follow-up session at least 6 months after post-test (week 30).
  We will implement a non-trained version of the n-back task, and for those in the multi-component training group, we will also include non-trained versions of each of the trained tasks. Dependent variables: Speed and accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Seitz, PhD, Principal Investigator — Northeastern University; Susanne Jaeggi, PhD, Principal Investigator — Northeastern University
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (anonymized).
Supporting Information: SAP, ICF
Time Frame: Data will be available persistently at the conclusion of the study.
Access Criteria: There are no access criteria.